CLINICAL TRIAL: NCT00214110
Title: Phase 2 Randomized Single-blind Escalating Dose Response Clinical Trial of Tamoxifen Therapy on Mean Percent Predicted Isometric Strength in Amyotrophic Lateral Sclerosis [ALS]
Brief Title: Tamoxifen Therapy in Amyotrophic Lateral Sclerosis [ALS]
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 2000-486
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2015-10-05 (Estimated); Status verified 2008-08

CONDITIONS: Amyotrophic Lateral Sclerosis (ALS)
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Tamoxifen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Tamoxifen

SUMMARY:
This is a single-center, phase 2 randomized clinical trial of tamoxifen on mean percent predicted isometric muscle strength in patients with amyotrophic lateral sclerosis (ALS). The purpose is to determine whether the triphenylethylenetamoxifen, used as adjuvant therapy in the treatment of breast cancer, can delay the loss of isometric muscle strength in ALS patients.

ELIGIBILITY:
Inclusion Criteria:

* clinically probable-laboratory supported, clinically probable, or clinically definite amyotrophic lateral sclerosis

Exclusion Criteria:

* Allergic or idiosyncratic response to tamoxifen.
* Other active neurologic diseases that may produce weakness, sensory loss, or autonomic symptoms.
* Psychiatric, psychological, or behavioral symptoms that would interfere with the subject's ability to participate in the trial.
* Clinically significant cardiac, pulmonary, gastrointestinal, hematologic, or endocrine (poorly controlled insulin-dependent diabetes mellitus or hyperthyroidism) disease that may confound interpretation of the study results.
* Previous kidney or pancreas transplants.
* Significant hepatic or renal disease (AST > 5 times normal, serum creatinine > 2.0 mg/dL for males or > 1.8 mg/dL for females).

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2001-01; Study Completion 2005-01 (Actual)

PRIMARY OUTCOMES:
Stability at 6, 12, 18 and 24 months on of the patient's mean percent predicted arm strength

SECONDARY OUTCOMES:
Vital capacity, raw liters and percent predicted, compared with baseline measured at 3 month intervals.
Individual arm and leg muscle mean percent predicted isometric strength compared with baseline measured at 3 month intervals.
Bulbar, Breathing, arm and leg subscores of ALS Functional Rating Scale - Revised [ALS-FRS-R] compared with baseline measured at 3 month intervals.
Total ALS Functional Rating Scale [ALS-FRS-R] compared with baseline measured at 3 month intervals.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin R Brooks, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States